CLINICAL TRIAL: NCT05057117
Title: Longevity of Microwave Thermolysis and Botulinum Toxin A for Treatment of Axillary Hyperhidrosis: a Randomized Intra-individual Trial
Brief Title: Longevity of Microwave Thermolysis and Botulinum Toxin A for Treatment of Axillary Hyperhidrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merete Haedersdal (Other)
Responsible Party: Sponsor-Investigator, Merete Haedersdal, Consultant in Dermatology, Clinical Professor, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MWT-BTXA; 2021-000877-10 (EudraCT Number); H-21013548 (Other: The Regional Health Research Ethics Committee)
Record Dates: First submitted 2021-09-07; First posted 2021-09-27 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Hyperhidrosis Primary Focal Axilla
Keywords: Axillary hyperhidrosis; Microwave thermolysis; Botulinum toxin A
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: A single-center, prospective, randomized, intra-individual, clinical trial comparing longterm efficacy of two treatments for axillary hyperhidrosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin A (Active Comparator): One treatment with standard dosage (50-100 units) of botulinum toxin A in one axilla
  Interventions: Drug: Botulinum toxin A
- Microwave thermolysis (Active Comparator): One standard treatment (energy level 5) with microwave thermolysis in one axilla
  Interventions: Device: Microwave thermolysis

INTERVENTIONS:
Device: Microwave thermolysis — Baseline treatment with microwave thermolysis in one axilla and botulinum toxin A in the contralateral axilla, as allocated by randomization
  Other Names: miraDry
  Arms: Microwave thermolysis
Drug: Botulinum toxin A — Baseline treatment with microwave thermolysis in one axilla and botulinum toxin A in the contralateral axilla, as allocated by randomization
  Other Names: Botox
  Arms: Botulinum toxin A

SUMMARY:
This trial aims is to assess and compare treatment effect of microwave thermolysis and botulinum toxin A for axillary hyperhidrosis with focus on longevity. The investigators also aim to assess patient satisfaction and adverse reactions in relation to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent
2. Subject is 18 years of age or older
3. A unilateral HDSS score of 3 or 4 for each axilla
4. A gravimetric measurement of at least 50 mg/5 min for women and 100 mg/5 min for men in at least one axilla. The contralateral axilla should not be below 40 mg (women) and 80 mg (men).
5. Women of childbearing potential must be confirmed not pregnant by a negative u-HCG prior to study treatment and must use a safe contraceptive method at baseline.

Exclusion Criteria:

1. Subjects with generalized hyperhidrosis
2. Medical condition or medications that may alter perspiration (e.g. metabolic, immunological or infectious diseases, antidepressants, opioids, adrenergic/cholinergic drugs)
3. Daily use of systemic or topical antibiotics and/or steroids in axillae at the time of inclusion
4. Topical treatments for axillary hyperhidrosis (anti-perspirants are allowed except for visit days)
5. Abnormal skin (e.g. rash, infection, dermatitis) in the axilla at the time of inclusion
6. Breast tissue in the axillae
7. Treatment with Isotretinoin within the past 6 months
8. Axillary laser or IPL treatment within the past 6 months
9. Botulinum toxin-injections in the axillae within the past 12 months prior to baseline
10. Known allergies to botulinum toxin, iodine, lidocaine or adrenaline
11. Prior axillary surgery
12. Limited motion in the shoulder joint or neurologic deficit in upper limb
13. History of diseases resulting in muscle weakness (ALS, Lou Gehrig's), dysphagia (Myasthenia Gravis or Lambert Eaton Syndrome) or respiratory compromise
14. Axillary lymph node enlargement or -removal or lymphedema in either upper limb
15. History of hidradenitis suppurativa or history of reoccurring infections/abscesses
16. History of breast cancer
17. Electronic device implant
18. If female; lactating, pregnant or planning on becoming pregnant during the study
19. Non-eligibility at the discretion of the investigator (e.g. non-compliance, unavailability or other reasons the subject is not believed to be able to comply with the clinical trial protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Subjective change in axillary sweat | Baseline - 6 months
  Unilateral sweat change from baseline to 6 months follow-up assessed by Hyperhidrosis Disease Severity Scale

SECONDARY OUTCOMES:
Objective change in axillary sweat | Baseline - 6 months
  Unilateral sweat change from baseline to 6 months follow-up assessed by gravimetric test
Patient Satisfaction | Baseline - 6 months - 12 months
  Unilateral patient satisfaction 6 and 12 months after treatments assessed on a 3-point Likert Scale (unsatisfied - neutral - satisfied)
Adverse reactions | Baseline - 12 months
  Unilateral evaluation of adverse reactions after treatments

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD PhD DMSc, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Department of Dermatology, Bispebjerg Hospital, Copenhagen, Denmark